CLINICAL TRIAL: NCT02306538
Title: Evaluation of Myocardial Changes During BReast Adenocarcinoma Therapy to Detect Cardiotoxicity Earlier With MRI - The EMBRACE MRI Study
Brief Title: Evaluation of Myocardial Changes During BReast Adenocarcinoma Therapy to Detect Cardiotoxicity Earlier With MRI
Acronym: EMBRACE-MRI
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 13-6543C
Record Dates: First submitted 2014-11-11; First posted 2014-12-03 (Estimated); Last update posted 2023-02-14 (Actual); Status verified 2022-05

CONDITIONS: Breast Neoplasms
Keywords: edema; inflammation; scar; ejection fraction; volumes
MeSH Terms: conditions — Breast Neoplasms; Edema; Inflammation; Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodwork
Oversight: Data Monitoring Committee: No

SUMMARY:
Breast cancer is the most common cancer amongst Canadian women. 15-20% of early breast cancers have high levels of a protein called HER2 which is associated with worse survival. Treatment of these patients with anthracyclines followed by trastuzumab (which targets HER2) improves survival. Unfortunately, these medications together can cause heart muscle injury resulting in heart dysfunction or failure in about 14% and 3.6% of the patients, respectively. Once heart failure (HF) occurs, about 60% of patients will not live past 2 years. Studies have suggested that patients with heart injury caused by anthracyclines may be more likely to develop HF with addition of trastuzumab. Therefore tests to find early heart injury after anthracyclines may allow doctors to start heart protective medications with the hope of preventing HF. Also, animal and small patient studies have shown that an increase in the water levels of the heart muscle (edema) may be an early sign of heart injury from anthracyclines. Cardiac MRI is a unique technique that has been shown to detect edema in various heart diseases.

The investigators will test the theory that, in women receiving treatment for breast cancer, heart edema detected by MRI at the end of anthracyclines will identify patients who will later develop heart dysfunction. MRI studies with novel techniques will be done pre-therapy, after anthracyclines, during herceptin, and at end of all therapy. The investigators will compare patients with and without heart dysfunction to test if patients with heart dysfunction are more likely to have edema after anthracyclines. Ultimately the investigators hope to use cardiac MRI to identify high risk patients and study various heart protective medications to prevent HF. This will improve the personal health of cancer patients by allowing them to live free of heart disease after their cancer therapy. Ultimately at a population level this will allow doctors to provide care that can be uniquely designed for each patient based on their individual risk.

The first 136 patients enrolled are included in the first part of the study, named EMBRACE-MRI 1. Enrollment for this part of the study is complete.

The remaining 44 patients will be enrolled into EMBRACE-MRI 2, which includes slight differences in obtaining sequences in MRI imaging.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo treatment with one of the following regimens: (a) 5-fluorouracil, epirubicin, cyclophosphamide, followed by docetaxel and trastuzumab, (b) adriamycin, cyclophosphamide, followed by docetaxel and trastuzumab, (c) adriamycin-cyclophosphamide with weekly paclitaxel and trastuzumab, or (d) dose dense adriamycin and cyclophosphamide followed by dose dense paclitaxel and trastuzumab
* Able to tolerate five ~60 minute CMR examinations over 15 months
* Able to give informed consent

Exclusion Criteria:

* Life expectancy < 12 months
* Participating in a clinical trial of a new cancer drug
* Having received previous anthracycline
* History of myocardial infarction or previous heart failure
* Current unstable angina, persistent atrial fibrillation or other irregular rhythm, or a history of more than mild regurgitant or stenotic valvular heart disease
* Severely reduced renal function (GFR ≤ 30 milliliters/minute)
* General MRI contraindications
* Baseline LVEF <55% by echo
* echocardiography image quality inadequate for strain analysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women ≥18 years with stage I-III, HER2+ breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The presence of myocardial edema stratified by the presence or absence of conventionally defined cardiotoxicity (this is a binary outcome). | 2-15 months
  Myocardial edema is defined as an 8% increase in segmental T2 values measured in milliseconds in at least 2 myocardial segments at either of the 2 early time points. Cardiotoxicity is defined as Cardiac Magnetic Resonance Imaging (CMR) measured (1) ≥5% absolute reduction in Left Ventricular Ejection Fraction (LVEF) from baseline to an LVEF <55% with signs or symptoms of HF, OR (2) a ≥10% absolute reduction in LVEF from baseline to <55% without accompanying signs or symptoms at the time points when CMR is obtained OR (3) the same amount of reduction in LVEF as above, identified by echo at any time point (done every 3 months) and confirmed by CMR at that time.

SECONDARY OUTCOMES:
The presence of edema stratified by the presence or absence of any drop in LVEF ≥5% by CMR by end of therapy (this is a binary outcome). | 2-15 months
  Please see definition for edema above

CONTACTS AND LOCATIONS:
Overall Officials: Paaladinesh Thavendiranathan, MD, Principal Investigator — University Health Network, Toronto; Bernd Wintersperger, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang F, Rankin K, Sooriyakanthan M, Signorile M, Steve Fan CP, Thampinathan B, Marwick TH, Osataphan N, Yu C, Koch CA, Amir E, Hanneman K, Abdel-Qadir H, Wintersperger BJ, Thavendiranathan P. Phenotypes of Myocardial Dysfunction on Serial Echocardiography and CMR in Women With Early-Stage Breast Cancer. JACC Cardiovasc Imaging. 2025 May;18(5):540-553. doi: 10.1016/j.jcmg.2024.12.010. Epub 2025 Mar 19. PMID 40117396
- [Derived] Calvillo-Arguelles O, Thampinathan B, Somerset E, Shalmon T, Amir E, Steve Fan CP, Moon S, Abdel-Qadir H, Thevakumaran Y, Day J, Woo A, Wintersperger BJ, Marwick TH, Thavendiranathan P. Diagnostic and Prognostic Value of Myocardial Work Indices for Identification of Cancer Therapy-Related Cardiotoxicity. JACC Cardiovasc Imaging. 2022 Aug;15(8):1361-1376. doi: 10.1016/j.jcmg.2022.02.027. Epub 2022 May 11. PMID 35926895
- [Derived] Esmaeilzadeh M, Urzua Fresno CM, Somerset E, Shalmon T, Amir E, Fan CS, Brezden-Masley C, Thampinathan B, Thevakumaran Y, Yared K, Koch CA, Abdel-Qadir H, Woo A, Yip P, Marwick TH, Chan R, Wintersperger BJ, Thavendiranathan P. A Combined Echocardiography Approach for the Diagnosis of Cancer Therapy-Related Cardiac Dysfunction in Women With Early-Stage Breast Cancer. JAMA Cardiol. 2022 Mar 1;7(3):330-340. doi: 10.1001/jamacardio.2021.5881. PMID 35138325
- [Derived] Houbois CP, Nolan M, Somerset E, Shalmon T, Esmaeilzadeh M, Lamacie MM, Amir E, Brezden-Masley C, Koch CA, Thevakumaran Y, Yan AT, Marwick TH, Wintersperger BJ, Thavendiranathan P. Serial Cardiovascular Magnetic Resonance Strain Measurements to Identify Cardiotoxicity in Breast Cancer: Comparison With Echocardiography. JACC Cardiovasc Imaging. 2021 May;14(5):962-974. doi: 10.1016/j.jcmg.2020.09.039. Epub 2020 Nov 25. PMID 33248962